CLINICAL TRIAL: NCT00928525
Title: Open-label Trial of Imatinib in Patients With Desmoid Tumor and Chondrosarcoma
Brief Title: Imatinib in Patients With Desmoid Tumor and Chondrosarcoma
Acronym: Basket 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571 Basket 1; EudraCT Number: 2006-006446-33
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2018-12

CONDITIONS: Advanced Desmoid Tumor; Advanced Chondrosarcoma
Keywords: PDGFr alpha; PDGFr beta; KIT
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib Mesylate (Experimental): Patients affected by Desmoid Tumor and Chondrosarcoma will receive Imatinib Mesylate 800 mg p.o./day (400 mg b.i.d.) for a maximum of 24 months
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — 800 mg p.o./day (400 mg b.i.d.) for a maximum of 24 months

SUMMARY:
The purpose of this study is to determine whether Imatinib Mesylate is active in diseases - such as Desmoid Tumor and Chondrosarcoma - expressing the receptor for the platelet-derived growth factor (PDGF) both in its isoform alpha and beta

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of DT or CDS.
* Biomolecular or immunohistochemical evidence of Imatinib mesylate target (KIT, PDGFRα PDGFRβ activation and/or presence of PDGFα or PDGFβ)
* Measurable or evaluable disease
* Surgical resection of local disease unfeasible radically (or unaccepted by the patient, or amenable to become less demolitive, or easier, or likely more feasible, after cytoreduction) and/or metastatic disease.
* ECOG Performance status 0, 1, 2 or 3
* Adequate bone marrow, liver and renal function
* Female patients of child-bearing potential must have negative pregnancy test.
* Male and female patients of reproductive potential must agree to employ an effective method of birth control throughout the study.
* Written, voluntary, informed consent.

Exclusion Criteria:

* Previous treatment with any other investigational or not investigational agents within 28 days of first day of study drug dosing
* Other primary malignancy with <5 years clinically assessed disease-free interval, except basal cell skin cancer or cervical carcinoma in situ.
* Grade III/IV cardiac problems as defined by the New York Heart Association Criteria
* Severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection)
* Known brain metastasis.
* Known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
* Known diagnosis of human immunodeficiency virus (HIV) infection.
* Previous radiotherapy to >/=25% of the bone marrow or within the previous 2 months on target lesion.
* Major surgery within 2 weeks prior to study entry.
* Expected non-compliance to medical regimens (e.g. psychiatric diseases).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Tumor response will be evaluated by different imaging techniques | every three months

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Centro di Riferimento Oncologico - Unit of Medical Oncology, Aviano, Pordenone
  - I.R.C.C. - Unit of Medical Oncology, Candiolo, Torino
  - Istituti Ortopedici Rizzoli - Unit of chemotherapy of Muscoloskeletal Tumors, Bologna
  - Policlinico S.Orsola Malpighi - Unit of Medical Oncology, Bologna
  - Istituto Nazionale Tumori - Unit of Medical Oncology, Milan
  - Istituto Nazionale Tumori Regina Elena - Unit of Medical Oncology I, Roma
  - Ospedale Gradenigo - Unit of Medical Oncology, Torino